CLINICAL TRIAL: NCT05611567
Title: A Feasibility Study Examing the Primary Obesity Surgery Endoluminal (POSE) 2.0 Procedure for the Management of Non-alcoholic Fatty Liver Disease
Brief Title: Endoscopic Gastric Plication Using the POSE2.0 Technique for Management of Fatty Liver Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emirates Health Services (EHS) (Other Government)
Collaborators: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Mariam Salem Alkhatry, Chair of Gastroenterology, Emirates Health Services (EHS)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DD/CTMD2/019/2019
Record Dates: First submitted 2022-10-27; First posted 2022-11-10 (Actual); Last update posted 2022-11-10 (Actual); Status verified 2022-11

CONDITIONS: Non-Alcoholic Fatty Liver Disease; Obesity
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Obesity | interventions — Behavior Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- POSE2.0 (Experimental): This is the arm that got the POSE2.0 procedure. The POSE 2.0 involves full-thickness plications by suture anchor pairs that shorten and tabularize the stomach along its greater curvature. The POSE 2.0 procedure was carried out using the Incisionless Operating Platform (USGI Medical, San Clemente, CA). This device is registered and commercially available in the United Arab Emirates for the management of obesity.
  Interventions: Procedure: POSE2.0 procedure; Behavioral: Life style and behavioral intervention
- Life style and behavioral intervention (Active Comparator): This is the comparator arm that received lifestyle modification alone for weight loss and NAFLD management (representing the comparative control group). This group underwent the same lifestyle program and clinical follow-up as the POSE2.0, but under a parallel standard clinical care pathway, which is the standard clinical pathway in the hospital this study was conducted in.
  Interventions: Behavioral: Life style and behavioral intervention

INTERVENTIONS:
Procedure: POSE2.0 procedure — The POSE 2.0 involves full-thickness plications by suture anchor pairs that shorten and tabularize the stomach along its greater curvature. The POSE 2.0 procedure was carried out using the Incisionless Operating Platform (USGI Medical, San Clemente, CA)
  Arms: POSE2.0
Behavioral: Life style and behavioral intervention — The intervention focuses on caloric restriction diet, physical activity, and behavioral modification targeted toward weight loss and administered by a health care professional months for the 12 months duration of the study.

SUMMARY:
Primary Obesity Surgery Endoluminal 2.0, or POSE 2.0, (USGI Medical, San Clemente, CA) creates full-thickness plications of gastric tissue endoscopically to shorten the stomach and narrow its aperture for weight loss in patients with obesity. Adults with obesity and non-alcoholic NAFLD were allocated based on preference and motivation to undergo the POSE 2.0 procedure with lifestyle modification or lifestyle modification alone to study the impact of the POSE2.0 procedures on NAFLD parameters and metabolic profile. Co-primary endpoints included improvement in controlled attenuation parameter (CAP) and resolution of hepatic steatosis at 12 months. Secondary endpoints included total body weight loss (TBWL), change in serum measures of hepatic steatosis and insulin resistance, and device safety.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated informed consent form.
2. Subject agrees to be compliant with study requirements and adhere to post-operative dietary & exercise recommendations for the duration of the study.
3. Subjects age >=18 years old.
4. Hepatic steatosis from NAFLD, as defined by a controlled attenuation parameter ≥ 280 dB/m without alternate cause of liver disease measured by a Fibroscan XL.
5. Body Mass Index ≥ 30kg/m2
6. If female, be either post-menopausal, surgically sterile, or agree to practice birth control during year of study and have negative serum HCG at screening/baseline.
7. Absence of current severe systemic disease (including, but not limited to: coronary artery disease, chronic obstructive pulmonary disease, congestive heart failure, cancer, and chronic renal disease).
8. Agrees not to undergo any additional weight loss interventional procedures or liposuction for 12 months following study enrollment.
9. Have not taken any prescription or over-the-counter weight loss medications OR those that can suppress appetite/induce weight loss for at least 6 months and agrees not to utilize for 12 months following study enrollment (including all stimulant medication).
10. Subjects must be willing to possibly forego any future weight loss procedures (i.e. Vertical Sleeve Gastrectomy) given the unknown long-term effects.
11. Residing within a reasonable distance from the Investigator's treating office (~50 miles) and willing and able to travel to the Investigator's office to complete all routine follow-up visits.

Exclusion Criteria:

1. History of (or intra-operative evidence of) prior bariatric, gastric or esophageal surgery.
2. Esophageal stricture or other anatomy and/or condition that could preclude passage of endoluminal instruments or procedure execution.
3. Moderate gastro-esophageal reflux disease (GERD), defined as symptoms that cause subject severe discomfort, compromise performance of daily activities, and/or condition is not entirely controlled with drug therapy.
4. Large hiatal hernia (>3 cm) by history or as determined by pre-enrollment endoscopy.
5. Pancreatic insufficiency/disease.
6. History of gastroparesis or symptoms that would be suggestive of gastroparesis or generalized dysmotility (e.g. esophago-gastric motility issues and lower esophageal sphincter abnormalities).
7. Pregnancy or plans of pregnancy in the next 12 months.
8. History of a known diagnosis or pre-existing symptom of rheumatoid arthritis, scleroderma, system lupus, or other autoimmune connective tissue disorder.
9. Immunosuppressive medications or systemic steroids (i.e., oral prednisone) within 6 months of Visit 1. Intranasal/inhaled steroids are acceptable.
10. Unable or unwilling to avoid use of aspirin and/or non-steroidal anti-inflammatory drugs (NSAIDs), or other medications known to be gastric irritants beginning two weeks prior to enrollment and throughout the entire study.
11. History of inflammatory disease of the GI tract; coagulation disorders; hepatic insufficiency or cirrhosis.
12. Active gastric erosion, lesion, or gastric/duodenal ulcer.
13. History of or current platelet or coagulation dysfunction, such as hemophilia.
14. History or present use of insulin or insulin derivatives for treatment of diabetes.
15. Type II Diabetes Mellitus (as defined by HgbA1c >6.5%) for greater than 11 years at the time of enrollment.
16. If smoker, plans to quit smoking in the year after enrollment.
17. Portal hypertension and/or varices.
18. Patient has a history of drug or alcohol abuse or positive at screening for drugs of abuse.
19. Present or history of psychosis, bipolar disease, or obsessive-compulsive disorder after pre-enrollment history and medical /psychological assessment.
20. Beck Depression Inventory (Short) Score ≥ 12 and/or uncontrolled depression after pre-enrollment psychological and medical assessment. 1
21. Patient score >2 in any of the 9 identified symptoms on the Gastroparesis Cardinal Symptom Index (GCSI)
22. Non-ambulatory or has significant impairment of mobility (i.e. cannot ambulate for 30 minutes).
23. Known hormonal or genetic cause for obesity including untreated hypothyroidism (TSH >5.0 U/ml).
24. Participating in another clinical study.
25. Subjects with a personal history of allergic/anaphylactic reactions including hypersensitivity to the drugs or materials that will be utilized in the study procedure.
26. Physician's assessment that the subject is not an appropriate candidate.

    -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2020-01-20 (Actual); Primary Completion 2022-03-15 (Actual); Study Completion 2022-09-01 (Actual)

PRIMARY OUTCOMES:
Change in controlled attenuation parameter (CAP) | 12 months
  Measured by Fibroscan XL
Change in liver stiffness | 12 months
  Measured by Fibroscan XL

SECONDARY OUTCOMES:
Percent resolution of hepatic steatosis at 12 months | 12 months
  Measured by fibroscan XL

OTHER OUTCOMES:
Change in total body weight loss (TBWL) in each arm | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Obaidulla Hospital, Emirates Health Services, Ministry of Health, United Arab Emirates, Ras al-Khaimah, United Arab Emirates

IPD SHARING:
Plan to Share IPD: Yes
Select IPD could be shared after approval of the UAE Ministry of Health and after signing a data-sharing agreement.
Supporting Information: Study Protocol, CSR, Analytic Code
Time Frame: Data is available for the next 2 years.

REFERENCES:
- [Derived] AlKhatry M, Rapaka B, Maselli DB, Abboud DM, Brunaldi VO, Mahmoud T, Ghazi R, Abdul Razzak F, Gala K, Joudah I, Housen F, Al Qadi S, Vargas EJ, Storm AC, Abu Dayyeh BK. Improvements in hepatic steatosis, obesity, and insulin resistance in adults with nonalcoholic fatty liver disease after the primary obesity surgery endoluminal 2.0 procedure. Endoscopy. 2023 Nov;55(11):1028-1034. doi: 10.1055/a-2117-6274. Epub 2023 Jun 26. PMID 37364600